CLINICAL TRIAL: NCT04363151
Title: Management of Liver Hydatid Cysts: A Retrospective Analysis of 293 Cases From Southern Iran
Brief Title: The Current Study Aimed to Evaluate the Therapeutic Features and Complications of Liver Hydatid Cyst in Patients Who Underwent Surgery for CE in Fars Province, Southern Iran.
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bahador Sarkari, Pronciple investigator, Shiraz University of Medical Sciences
Other Study IDs: 94-01-01-9212
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Patients Who Underwent Surgury for Hydatid Cyst
Keywords: Hydatid cyst, Surgery, hospital record
MeSH Terms: conditions — Echinococcosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hydatid cyst patients: patients who underwent surgery for liver hydatid cyst from 2004 to 2018 in two major university-affiliated hospitals in Fars Province, southern Iran
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention.

SUMMARY:
The current study aimed to evaluate the therapeutic features and complications of liver hydatid cyst in patients who underwent surgery for CE in Fars province, southern Iran.

A total of 293 patients who underwent surgery for liver hydatid cyst from 2004 to 2018 in Fars Province, southern Iran, were retrospectively evaluated. The clinical records of patients were reviewed and the demographic and clinical characteristics of each patient were assessed.

DETAILED DESCRIPTION:
Fars province with the capital of Shiraz in one of the thirty-one provinces of Iran located in the southwest part of the country with a population of more than 4.6 million people of which 67.6% living in urban areas, 32.2% in rural areas and 0.3% live as nomad tribes. The average temperature of Fars province is 17.8 °C, ranging between 4.7 °C and 29.2 °C and the annual rainfall is 261mm. Animal farming and agriculture are of great importance as they are considered as two main economic bases of this province. This type of livelihood has facilitated the presence of some of the zoonotic diseases such as CE and toxocariasis and leishmaniasis.

Data Collection Hospital records of a total of 293 patients who underwent surgery for liver hydatid cyst from 2004 to 2018 in two major university-affiliated hospitals in Fars Province, southern Iran, were retrospectively evaluated. In all cases, the preliminary diagnosis of hydatid cyst has been confirmed by postoperative pathological findings. So, the inclusion criterion of operation with the diagnosis of CE was considered while reviewing the records.

Information such as age, sex, presenting signs and symptoms of hydatid cyst, number and the specific location of cystic structures, history of relapse, reoperation, characteristics of the cyst (calcification, puss discharge, multicystic, multiloculated, daughter cyst, rupture, inflammation, superimposed infection, and septation), early postoperative complications, diagnostic procedures such as ultrasound scanning, computed tomography, X-rays, pathology reports, lab data, operation information and, drug therapy were extracted from the hospital records of each patient. The surgical procedure used for the patients, radical or conservative, was noted.

ELIGIBILITY:
Inclusion Criteria:

Having a surgery due to Hydatid cyst

Exclusion Criteria:

Surgeries other than hydatid cyst.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 293 patients who underwent surgery for liver hydatid cyst from 2004 to 2018 in two major university-affiliated hospitals in Fars Province, southern Iran.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2004-01-15 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Demographic Information as well as patients clinical data were extracted from the hospital records of each patient. | 2004 to 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
The individuals' data will not be shared with other researchers, as there is no need to do so.